CLINICAL TRIAL: NCT07072676
Title: The Use of Assistive Gait Devices Can Reduce the Risk of Falls in Patients With Neuromuscular Diseases Following a Training Period.
Acronym: Risk of fall
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Marko Mijic, Principal Investigator, LMU Klinikum
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-0252; 25-0252 (Registry Identifier: ETHICS COMMITTEE AT THE LMU MUNICH)
Record Dates: First submitted 2025-06-27; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Inclusion Body Myositis; Myotonic Dystrophy 1; Myotonic Dystrophy 2; Facio-Scapulo-Humeral Dystrophy; Limb Girdle Muscular Dystrophies; Pompe Disease (Infantile-Onset); Myasthaenia Gravis; Lambert Eaton (LEMS); Spinal Muscular Atrophy (SMA); Guillain Barré Syndrome; Chronic Inflammatory Demyelinating Polyneuropathy; Friedreich Ataxia; Hereditary Motor and Sensory Neuropathies
Keywords: assistive gait device, neuromuscular diseases
MeSH Terms: conditions — Myositis, Inclusion Body; Myotonic Dystrophy; Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies, Limb-Girdle; Glycogen Storage Disease Type II; Lambert-Eaton Myasthenic Syndrome; Muscular Atrophy, Spinal; Guillain-Barre Syndrome; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Friedreich Ataxia; Hereditary Sensory and Motor Neuropathy; Neuromuscular Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A study protocol was developed with two cohorts that underwent a one-week pre-post intervention with gait assistive devices. The first group consisted of patients (n= 15) requiring orthopaedic support: Knee and/or ankle foot orthoses and orthopaedic shoes; the second group (n= 15) consists of patients requiring mobility aids: Forearm crutches, rollators and walking aids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention period (No Intervention): One week without therapy with asssisitive gait devices. During this week, patients undergoing inpatient rehabilitation receive standard therapy for neuromuscular disorders.
- Intervention period (Experimental): One week therapy with assisitve gait devices.
  Interventions: Device: Assistive gait devices combined with physiotherapy

INTERVENTIONS:
Device: Assistive gait devices combined with physiotherapy — During the intervenation week, the patient undergoes 12 hours/week of gait training, fall prevention, balance group and physiotherapy as part of their inpatient rehabilitation programme. The individual sessions last 30 minutes each.
  Arms: Intervention period

SUMMARY:
The planned project is an intervention study to assess the risk of falling after adaptation of an assistive gait devices in patients with the following neuromuscular diseases: Inclusion body myositis, myotonic dystrophy, limb girdle and facioscapulohumeral muscular dystrophies, Pompe disease, Lambert-Eaton syndrome, myasthenia gravis, spinal muscular atrophy, Guillain-Barré syndrome, chronic inflammatory demyelinating polyradiculoneuropathy, Friedreich's ataxia and hereditary motor and sensory neuropathy.

The primary aim is to assess the risk of falling after a suitable assistive gait device has been provided with an adaptation phase through training. The data should help to improve the provision of aids for patients with neuromuscular diseases. This should have a positive effect on the risk of falling and thus improve quality of life and reduce mortality and morbidity. To achieve these goals, a one-week intervention with training sessions on handling, balance and coordination as well as fall prevention will becarried out after the patient has been fitted with a suitable assistive gait device.

The interventions will be embedded in the inpatient rehabilitation programme. The functional gait and balance tests 'Timed Up and Go', '10 metre walk test', '6-minute walk test' and 'Dynamic Gait Index' will be recorded additionally.

The Falls Efficacy Scale International questionnaire will be utilised to evaluate the risk of falling, while the Quebec User Evaluation of Satisfaction with Assistive Technology questionnaire will be employed to ascertain satisfaction with the assistive devices. The study is scheduled to run for a period of 14 days, during which participants will undergo three functional walking and balance tests. As part of the inpatient rehabilitation programme, participants will undergo a week-long period of rehabilitation without assistive technology, followed by a subsequent week of rehabilitation with adapted assistive technology.

ELIGIBILITY:
Inclusion Criteria:

* The Patients with sufficient cognitive and communicative abilities,
* The Patients with confirmed by the genetic report and/or the final clinical diagnosis.

Exclusion Criteria:

* The Patients scored more than 23 points on the falls efficacy Scale-International
* The Patients are unable to walk at least ten metres without assistance,
* The patient had knee, hip or back surgery in the last three months.
* Patients suffering from polyneuropathy without a diagnosis of inflammatory autoimmune neuropathy.

Ages: 65 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test | At Day 1, end of pre-intervention period Day 7, and at the end of post-intervation period Day 14.
  The aim of this test is to walk as far as possible for 6 minutes.
Timed Up and Go (TUG) | At Day 1, end of pre-intervention period Day 7, and at the end of post-intervation period Day 14.
  The TUG test measures the time it takes to stand up from a chair, walk three metres, turn around and sit back down on the same chair.
10 meter walk test | At Day 1, end of pre-intervention period Day 7, and at the end of post-intervation period Day 14.
  Walking at maximum speed is measured in a long, flat-surface corridor of 10 meters, with a standing start and a "flying" finish 2.5 meters beyond the 10-meter mark.
Dynamic Gait Index | At Day 1, end of pre-intervention period Day 7, and at the end of post-intervation period Day 14.
  Dynamic Gait Index tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions. It is a useful test in individuals with vestibular and balance problems and those at risk of falls.

SECONDARY OUTCOMES:
The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) | At the end of post-intervention period, Day 14.
  The QUEST 2.0 evaluates a patient's satisfaction with various assistive technologies.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Park, Bad Feilnbach, Reithofpark, Bad Feilnbach, Germany

IPD SHARING:
Plan to Share IPD: No
In accordance with the guidelines of the Ethics Committee.

REFERENCES:
- [Background] Dias N, Kempen GI, Todd CJ, Beyer N, Freiberger E, Piot-Ziegler C, Yardley L, Hauer K. [The German version of the Falls Efficacy Scale-International Version (FES-I)]. Z Gerontol Geriatr. 2006 Aug;39(4):297-300. doi: 10.1007/s00391-006-0400-8. German. PMID 16900450
- [Background] Waterval NFJ, Brehm MA, Altmann VC, Koopman FS, Den Boer JJ, Harlaar J, Nollet F. Stiffness-Optimized Ankle-Foot Orthoses Improve Walking Energy Cost Compared to Conventional Orthoses in Neuromuscular Disorders: A Prospective Uncontrolled Intervention Study. IEEE Trans Neural Syst Rehabil Eng. 2020 Oct;28(10):2296-2304. doi: 10.1109/TNSRE.2020.3018786. Epub 2020 Aug 24. PMID 32833637
- [Background] Ounpuu S, Garibay E, Acsadi G, Brimacombe M, Pierz K. The impact of orthoses on gait in children with Charcot-Marie-Tooth disease. Gait Posture. 2021 Mar;85:198-204. doi: 10.1016/j.gaitpost.2021.02.005. Epub 2021 Feb 12. PMID 33610823
- [Background] Mijic M, Wirner-Piotrowski C, Jung A, Gutschmidt K, Arndt M, Garcia-Angarita N, Wenninger S, Young P, Schoser B. The assistive gait devices and their implementation in activities of daily living for patients with neuromuscular disease: A systematic review and meta-analysis. J Neuromuscul Dis. 2026 Jan;13(1):53-76. doi: 10.1177/22143602241289216. Epub 2024 Dec 8. PMID 39973408
- [Background] Dharmadasa T, Matamala JM, Huynh W, Zoing MC, Kiernan MC. Motor neurone disease. Handb Clin Neurol. 2018;159:345-357. doi: 10.1016/B978-0-444-63916-5.00022-7. PMID 30482326
- [Background] Atalaia A, Thompson R, Corvo A, Carmody L, Piscia D, Matalonga L, Macaya A, Lochmuller A, Fontaine B, Zurek B, Hernandez-Ferrer C, Reinhard C, Gomez-Andres D, Desaphy JF, Schon K, Lohmann K, Jennings MJ, Synofzik M, Riess O, Yaou RB, Evangelista T, Ratnaike T, Bros-Facer V, Gumus G, Horvath R, Chinnery P, Laurie S, Graessner H, Robinson P, Lochmuller H, Beltran S, Bonne G. A guide to writing systematic reviews of rare disease treatments to generate FAIR-compliant datasets: building a Treatabolome. Orphanet J Rare Dis. 2020 Aug 12;15(1):206. doi: 10.1186/s13023-020-01493-7. PMID 32787960
- See also: Related Info — https://www.lmu-klinikum.de/friedrich-baur-institut